CLINICAL TRIAL: NCT03682978
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Arbaclofen Administered for the Treatment of Social Function in Children and Adolescents With Autism Spectrum Disorders
Brief Title: Arbaclofen in Children and Adolescents With ASD
Acronym: AIMS2-CT1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celso Arango, MD, PhD (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIMS2-CT-01; 2018-000942-21 (EudraCT Number)
Record Dates: First submitted 2018-09-07; First posted 2018-09-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Autism Spectrum Disorder
Keywords: Arbaclofen; Placebo-Controlled; Randomized; Double-Blind; Social Function; Efficacy; Safety; Tolerability; Children; Adolescents; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Social Adjustment | interventions — arbaclofen placarbil; Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AIMS2-CT-01 is a double-blind study where participants and parent(s)/legal guardians as well as research staff will be unaware of the treatment allocation, with the exception of a dedicated unblinded pharmacist at each individual site. Blinding of the remainder of the study team members will be maintained by utilizing identical tablets, blistercards and boxes containing either Arbaclofen or placebo. Unblinded study drug and placebo supplies will be stocked at each study site pharmacy. An online randomization system will be used, by this unblinded pharmacist, to assign the study treatment. Based on the outcome of the randomisation, the pharmacist prepares the boxes containing the applicable treatment and releases these (blinded) boxes to the investigator for dispensing to the patient. In order to maintain the study blind, the dosing regimen will be consistent whether participants are randomized to Arbaclofen or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arbaclofen (Experimental): Arbaclofen is provided as orally disintegrating tabs, round, white and beveled edges, at the following strengths: 5mg, 10mg, 15mg and 20mg.
  A flexible dose titration schedule will be utilized during the first 5 weeks of the Treatment Period. Dosing regimens will be stratified by age. The total up-titration to 15 mg TID or 20 mg TID, and dose adjustment period to the optimal dose will be 35 days. If a participant does not tolerate a dose increase, he or she should return to the previous dose level and must remain at the dose level for the remainder of the Treatment Period. No changes should be made to dosing after 5 weeks, unless for safety.
  5-11 years: Week 0 (BID) 5mg; Week 1 (BID) 5mg; Week 2 (TID) 10mg; Week 3 (TID) 10mg; Week 4-16 (TID) 15mg.
  12-17 years: Week 0 (QD) 5mg; Week 1 (BID) 10mg; Week 2 (BID) 10mg; Week 3 (TID) 15mg; Week 4-16 (TID) 20mg.
  Interventions: Drug: Arbaclofen
- Placebo (Placebo Comparator): Placebo tablets will have similar form, colour, smell and taste compared to the Arbaclofen tablets, and will be provided in non-distinguishable packaging.
  Dosage level is n/a.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arbaclofen — Arbaclofen tablet.
  Other Names: R-4-amino-3-(4-chlorophenyl) butanoic acid (R-baclofen); STX209; C10H12ClNO2
  Arms: Arbaclofen
Drug: Placebo — Placebo tablet.
  Other Names: Placebo (for Arbaclofen)
  Arms: Placebo

SUMMARY:
AIMS-2-CT-01 is a randomized, double-blind, placebo controlled, study to explore the efficacy, safety and tolerability of Arbaclofen administered to children and adolescents (ages 5-17) for the treatment of social adaptive function in participants with ASD. The effects of Arbaclofen on social function in children and adolescents with ASD will be evaluated in a randomized, placebo controlled, parallel-group study of 16 weeks duration. Subjects who meet protocol criteria will be randomly allocated to receive either Arbaclofen or placebo in a 1:1 ratio in the Treatment Period. There will be 7 recruiting sites and randomization will be stratified by site. A sample of 130 patients will be recruited. Blinding will be maintained by utilizing identical tablets containing either Arbaclofen or placebo.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a clinically and etiologically heterogeneous neurodevelopmental condition affecting approximately 1% of the population. The core symptoms of ASD are deficits in social communication and the presence of repetitive and restricted behaviours and interests, including sensory anomalies. Currently, there are no effective medical treatments for the core symptoms of ASD, and families frequently use costly non evidence based interventions. Developing drugs for ASD has been challenging because of a limited understanding of its underlying pathophysiology(ies), and difficulties modelling it in vitro and in vivo.

A recent study from EU-AIMS reported, for the first time in ASD, that differences in E-I balance can be 'shifted' using a GABA acting drug (riluzole), and that abnormalities in functional connectivity can be 'normalised' by targeting E-I, even in adults. This offers promise that drugs targeting specific parts of the GABA pathway may improve symptoms.

The aim of the investigator's project is to conduct a double-blind Randomized Control Trial (RCT) focused on GABA/glutamate equilibrium, to assess the efficacy of a drug that targets core and/or comorbid symptoms in ASD. Arbaclofen is a selective GABA-B receptor agonist and augments GABA-ergic activity, inhibits presynaptic release of glutamate, inhibits postsynaptic transmission, and modulates intracellular signalling. Through elevation of GABA-ergic inhibitory activity, Arbaclofen may act to alleviate ASD symptoms with social anxiety and emotional hyperarousal.

Hypothesis: Arbaclofen will be superior to placebo in improving social function as measured by the Vineland-3 social domain.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent

   1. Participants or their legal representative must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal participant care. Participants who do not have the capacity to consent will give developmentally appropriate assent.
   2. Participants must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing.
   3. The subject's parent/caregiver/LAR must be able to speak and understand the local language where the study is conducted sufficiently to understand the nature of the study and to allow for the completion of all study assessments. The same parent/caregiver/LAR must be capable of providing reliable information about the subject's condition, agree to oversee the administration of study drug, and accompany the subject to all clinic visits.
   4. Patient must be able to speak and understand the local language where the study is conducted sufficiently to understand the nature of the study and to allow for the completion of all study assessments.
2. Type of Participant and Target Disease Characteristics

   1. Diagnosis of an Autism Spectrum Disorder according to the DSM-5 criteria
   2. Complex language as defined in ADOS-2 to qualify for a Module 3 or 4.
   3. Current pharmacological treatment regimen affecting behaviour has been stable for at least 6 weeks prior to screening and is expected to be stable during the duration of the study
   4. Current psychotherapeutic/psychosocial interventions affecting behaviour stable for 3 months prior to screening and expected to be stable during the duration of the study (standard regular school breaks and/or annual teacher/classroom change do not qualify for intervention change).
   5. Subjects with a history of seizure disorder must currently be receiving stable treatment with anticonvulsant medication and must have been seizure free for 6 months prior to screening, or must be seizure free for 3 years prior to screening if not currently on a stable (>3 months) dose of antiepileptics.
3. Age, Residential and Reproductive Status

   1. Male or female participants 5 to 17 years of age at the time of providing consent, inclusive.
   2. Reside with the parent/carer who is interviewed for the Vineland.
   3. Negative pregnancy test for females of childbearing potential (subject has experienced onset of menses) within 24h prior to study treatment starts.
   4. Females of childbearing potential who are sexually active must agree to use a highly effective form of contraception (i.e., existing surgical sterilization, complete abstinence, or a combination of two effective forms of contraception, such as, for example, condoms plus hormonal treatment).
   5. Male participants with female partners of childbearing potential are eligible to participate if they agree to the following conditions:

      * Inform any and all partner(s) of their participation in a clinical drug study and the need to comply with contraception instructions as directed by the investigator.
      * Male participants are required to use a condom for study duration and until end of relevant systemic exposure defined as 7 months after the end of study treatment.
      * Female partners of males participating in the study to consider use of effective methods of contraception until the end of relevant systemic exposure, defined as 7 months after the end of treatment in the male participant.
      * Male participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse or use a male condom during each episode of penile penetration during the treatment and until 7 months after the end of study treatment.
      * Refrain from donating sperm for the duration of the study treatment and until 7 months after the end of study treatment.

Exclusion Criteria:

1. Medical Conditions

   a. Subjects with any condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being. This includes, but is not limited to impairment of renal function, evidence or history of malignancy or any significant haematological, endocrine, respiratory, hepatic, cardiovascular or gastrointestinal disease, including any clinically significant abnormalities on ECG. In general, any co-morbid conditions that may interact with study procedures.
2. Prior/Concomitant Therapy

   1. Subjects who are currently receiving treatment with racemic baclofen, vigabatrin, tiagabine, or riluzole or other GABA-related medications (e.g. gabapentin or pregabalin). Only occasional benzodiazepine (or derivative drugs) use (PM, i.e. at night) will be allowed.
   2. Subjects who are currently receiving pharmacologic treatment affecting behaviour (see concomitant medication section) need to have a stable dose during the 6 weeks prior to the screening visit and for the duration of the study.
   3. Participating in programs including non-pharmacologic educational, behavioural, and/or dietary interventions affecting behaviour, participation in these programs must have been continuous during the 3 months prior to screening and participants or their parent/caregiver/LAR may not electively initiate new or modify ongoing interventions for the duration of the study. Typical school vacations are not considered modifications of stable programming.
   4. Subjects who have taken another investigational drug within the last 30 days.
3. Physical and Laboratory Test Findings

   a. Patients with evidence of any significant hematological, endocrine, cardiovascular (including uncorrected symptomatic congenital heart disease), respiratory, renal, hepatic, or gastrointestinal disease, not including mild common pediatric diseases in these areas that are stable (e.g. mild asthma, constipation, etc.), as judged by the investigator.
4. Study Medication Related

   1. Subjects who are not able to take oral medications.
   2. Subjects who have a history of hypersensitivity to racemic baclofen.
   3. Subjects with rare hereditary problems of galactose intolerance, the lactase deficiency or glucose-galactose malabsorption should not take this medicine.
   4. Active peptic ulceration as Baclofen stimulates gastric acid secretion.
   5. Porphyria.
5. Other Exclusion Criteria

   1. Subjects who are currently engaged in illicit drug use or alcohol abuse, according to DSM-5 criteria.
   2. Subjects who have previously participated in a clinical trial of Arbaclofen.
   3. Women who are breastfeeding.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Effect of Arbaclofen vs. placebo on social function | Week 0 + Week 16
  Vineland-3 (socialization domain): The Vineland Adaptive Behavior Scales, Third Edition is designed to assess the personal and social functioning of handicapped and non-handicapped persons. It is a gold standard for the assessment of adaptive functioning. The Socialization domain is one of the 4 adaptive domains assessed by the comprehensive interview form. The other 3 adaptive domains are communication, daily living skills and motor skills. The Socialization domain has 3 subdomains: interpersonal relations, play and leisure and coping skills.

SECONDARY OUTCOMES:
Effect of Arbaclofen vs. placebo on measures of global function | Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  CGI-I: Clinical Global Impression - Improvement Scale is used to determine the patient's improvement in response to treatment.
Effect of Arbaclofen vs. placebo on measures of global function | Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  CGI-S: The Clinical Global Impression - Severity Scale is used to assess the impairment of neurobehavioral function in study subjects.
Effect of Arbaclofen vs. placebo on other adaptive domains | Week 0 + Week 16
  Vineland-3 (other adaptive domains): The Vineland Adaptive Behavior Scales, Third Edition, other adaptive domains: communication, daily living skills and motor skills.
Effect of Arbaclofen on measures of social abilities and responsiveness | Week -3
  ADOS-2: The Autism Diagnostic Observation Schedule, Version 2, will be used to assess autistic symptomatology.The ADOS-2 is a standardized protocol for the observation of social and communicative behaviour in children, adolescents, and adults who are suspected of having an ASD.
Effect of Arbaclofen on measures of social abilities and responsiveness through BOSCC | Week 0 + Week 16
  BOSCC: The Brief Observation of Social Communication Change will be used to to sensitively measure change of core autistic symptoms by observation of a semi-structured social interaction between a child and an examiner.
Effect of Arbaclofen on measures of social abilities and responsiveness through SRS-2-P | Week 0 + Week 16
  SRS-2-P: The Social Responsiveness Scale (parent version) measures the severity of social impairment in ASD.
Effect of Arbaclofen on measures of social abilities and responsiveness through SRS-2-T | Week 0 + Week 16
  SRS-2-T: The Social Responsiveness Scale (teacher version) measures the severity of social impairment in ASD.
Effect of Arbaclofen on measures of problem behaviours | Week 0 + Week 4 + Week 8 + Week 12 + Week 16
  ABC-C: This is the community version of the original residential version of the Aberrant Behaviour Checklist. It is designed to objectively identify five behaviour subscales through observation by the primary caregiver: irritability, lethargy, stereotypy, hyperactivity, and inappropriate speech.
Effect of Arbaclofen on measures of problem behaviours | Week 0 + Week 16
  CBCL: Child Behaviour Checklist is a caregiver report form identifying problem behaviour in children.
Effect of Arbaclofen on other measures of core symptoms | Week 0 + Week 4 + Week 8 + Week 12 + Week 16
  AIM: The Autism Impact Measure is designed to measure change in the core symptoms of autism.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with the SMURF | Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  SMURF: Safety Monitoring Uniform Research Form.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with the ESS-CHAD | Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  ESS-CHAD: The Epworth Sleepiness Scale for Children and Adolescents will be employed to evaluate sedation.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with the C-SSRS | Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  C-SSRS: The Columbia Suicide Severity Rating Scale is used to measure suicidality.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with a pulse rate measurement | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Vital signs: pulse
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with a body temperature measurement | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Vital signs: body temperature
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with a blood pressure measurement | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Vital signs: blood pressure
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed by measuring weight | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Weight: Weight (in kg) will be assessed with all outer wear and shoes removed.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed by measuring height | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Height: Height (in cm) will be assessed with all outer wear and shoes removed.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with the Tanner scale | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16 + Week 18
  Tanner stage
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with blood tests | Week -3 + Week 16
  Blood tests: CBC, serum chemistry, liver enzymes and renal function.
Safety and tolerability of Arbaclofen in children and adolescents with ASD as assessed with blood tests | Drug testing: Week -3 + Week 16, Pregnancy testing: Week -3 + Week 0 + Week 4 + Week 8 + Week 12 + Week 16
  Urine tests: basic urinalysis, toxics (amphetamines, benzodiazepines, barbiturates, marijuana/cannabis, cocaine, opioids (narcotics)) and pregnancy.
To explore the use and feasibility of digital biomarkers | Week -3 + Week 0 + Week 2 + Week 4 + Week 6 + Week 8 + Week 12 + Week 16
  To explore the use and feasibility of digital biomarkers as treatment-responsive measures of core and associated symptoms of ASD

OTHER OUTCOMES:
Explore whether P1 & N170 amplitude & latency as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  P1 & N170 amplitude & latency are assessed with a face ERP task.
Explore whether Alpha & Theta power (frontal) and Theta connectivity as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  Alpha & Theta power (frontal) and Theta connectivity are assessed by watching social and non-social videos.
Explore whether induced power at 10Hz & 40Hz as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  Induced power at 10Hz & 40Hz is assessed with an Auditory Steady State Response task.
Explore whether induced and evoked power at 6Hz & 10Hz as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  Induced and evoked power at 6Hz & 10Hz are assessed with a Visual Steady State Response task.
Explore whether P1, N1 amplitude and latency of standard stimuli and Mismatch Negativity (MMN) amplitude and latency as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  P1, N1 amplitude and latency of standard stimuli and Mismatch Negativity (MMN) amplitude and latency are assessed with a Visual Steady State Response task.
Explore whether Alpha & Theta power and connectivity as measures of electrophysiology (EEG) are associated with either response to treatment | Week 0 + Week 16
  Alpha & Theta power and connectivity are assessed with a Resting State task.
Explore the relationship between optional blood biomarkers (DNA) and safety, efficacy, and optimal dosing of Arbaclofen as assessed by the measurements specified in the previous outcome measures. | Week 0 + Week 16
  Optional blood biomarkers (DNA): The purpose of this repository is to allow future studies of the relationship between variation in DNA sequence with the safety, efficacy, and optimal dosing of Arbaclofen in the treatment of ASD.

CONTACTS AND LOCATIONS:
Overall Officials: Celso Arango, Prof., Study Chair — Hospital General Universitario Gregorio Marañón; Mara Parellada, Prof., Principal Investigator — Hospital General Universitario Gregorio Marañón; Richard Delorme, Prof., Principal Investigator — Hopital Universitaire Robert-Debre; Jeremy Parr, Prof., Principal Investigator — University of Newcastle Upon-Tyne; Mallika Punukollu, Dr., Principal Investigator — University of Glasgow; Andre Strydom, Prof., Principal Investigator — King's College London; Rosa Calvo, Dr., Principal Investigator — Hospital Clinic of Barcelona
Locations (7):
- Robert Debré Hospital, Paris, France
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Servicio de Psiquiatría del Niño y del Adolescente, Hospital General Universitario Gregorio Marañón, SERMAS, Madrid
  - University of Salamanca & Complejo asistencial de Zamora, Salamanca
- United Kingdom (3):
  - University of Glasgow, Glasgow
  - King's College London, London
  - University of Newcastle upon Tyne, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parellada M, San Jose Caceres A, Delorme R, Moscoso A, Moreno C, Calvo R, Canal-Bedia R, Franco Martin MA, Charman T, Strydom A, Parr JR, Urbiola Merino E, Burdeus-Olavarrieta M, Hernandez Jusdado P, Solis A, Lucas M, Sipos L, Gonzalez Navarro P, Blazquez A, Lazaro L, Tomas A, Humeau E, Antoun S, Cooke J, Megalogeni M, Liang H, de-Vena-Diez VB, Leonard H, White N, Wang P, Walton-Bowen K, Winter-van Rossum I, Murphy D, Arango C. Efficacy, safety, and tolerability of arbaclofen in Autistic children and adolescents, the AIMS-2-TRIALS-CT1: a randomized, double-blind, placebo-controlled phase II trial. EClinicalMedicine. 2026 Jan 22;92:103760. doi: 10.1016/j.eclinm.2026.103760. eCollection 2026 Feb. PMID 41631164
- [Derived] Parellada M, San Jose Caceres A, Palmer M, Delorme R, Jones EJH, Parr JR, Anagnostou E, Murphy DGM, Loth E, Wang PP, Charman T, Strydom A, Arango C. A Phase II Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Arbaclofen Administered for the Treatment of Social Function in Children and Adolescents With Autism Spectrum Disorders: Study Protocol for AIMS-2-TRIALS-CT1. Front Psychiatry. 2021 Aug 24;12:701729. doi: 10.3389/fpsyt.2021.701729. eCollection 2021. PMID 34504446
- See also: AIMS-2-TRIALS website — https://www.aims-2-trials.eu/